CLINICAL TRIAL: NCT05316311
Title: Implantation of CERENOVUS ENTERPRISE 2 Intracranial Stent in Patients With Severe Symptomatic Intracranial Atherosclerotic Stenosis: A Multicenter, Prospective and Single-Arm Study in China
Brief Title: A Study of Implantation of CRENEOUS ENTERPRISE 2 Intracranial Stent in Participants With Severe Symptomatic Intracranial Atherosclerotic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medos International SARL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNV202003; CNV202003 (Other: Medos International SARL)
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- CERENOVUS ENTERPRISE 2 Intracranial Stent (Experimental): Participants with severe symptomatic intracranial artery stenosis will be treated with CERENOVUS ENTERPRISE 2 Intracranial Stent.
  Interventions: Device: CERENOVUS ENTERPRISE 2 Intracranial Stent

INTERVENTIONS:
Device: CERENOVUS ENTERPRISE 2 Intracranial Stent — CERENOVUS ENTERPRISE 2 Intracranial Stent will be used to treat severe symptomatic intracranial artery stenosis.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of CERENOVUS ENTERPRISE 2 intracranial stent implantation in treatment of participants with severe symptomatic intracranial atherosclerotic stenosis.

ELIGIBILITY:
Inclusion Criteria:

Pre-procedure inclusion criteria

* Participants aged 22-80 years old
* All participants are required to meet at least one additional criteria (a-f) provided below to qualify for the study; (a) insulin dependent diabetes for at least 15 years; (b) at least 2 of the following atherosclerotic risk factors: hypertension (blood pressure [BP] greater than or equal to [>=] 140/90 or on antihypertensive therapy); dyslipidemia (low density lipoprotein [LDL] 130 milligrams per deciliter [mg/dl] or high density lipoprotein [HDL] less than [<] 40 mg/dl or fasting triglycerides >= 150 mg/dl or on lipid lowering therapy); smoking; abnormal glucose metabolism (fasting blood glucose >= 6.2 millimole per liter (mmol/L) or 2 hours postprandial blood glucose >= 7.8mmol/L); family history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, stroke, carotid endarterectomy or stenting, peripheral vascular surgery in parent or sibling who was <55 years of age for men or <65 for women at the time of the event ; (c) history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, carotid endarterectomy or stenting, or peripheral vascular surgery for atherosclerotic disease ; (d) any stenosis of an extracranial carotid or vertebral artery, another intracranial artery, subclavian artery, coronary artery, iliac or femoral artery, other lower or upper extremity artery, mesenteric artery, or renal artery that was documented by non-invasive vascular imaging or catheter angiography and is considered atherosclerotic ; (e) Aortic arch atheroma or atherosclerotic aortic aneurysm documented by non-invasive vascular imaging or catheter angiography ; (f) High resolution magnetic resonance imaging (MRI) imaging confirmed the presence of atherosclerotic plaques in the target arterial stenosis
* Participants with symptomatic intracranial atherosclerotic stenosis who is receiving medical treatment (that is, receiving at least one antithrombotic medication and vascular risk factor management) but still had recurrent (2 or more) ischemic strokes during the medical treatment period within past year
* Vascular diameter proximal to the stenosis must be measured at 2.0-4.0 millimeters (mm)
* Modified Rankin Scale (mRS) <= 2
* Stenosis of 70%-99% on non-invasive vascular imaging or digital subtraction angiography (DSA), with normal distal vessel
* Participant is willing and able to return for all follow-up visits required by the protocol
* Participants understand the purpose and requirements of the study and have signed an informed consent form Intra procedure
* Stenosis of 70 percent (%) -99% on digital subtraction angiography (DSA), with normal distal vessel

Exclusion Criteria:

* Participant underwent an acute ischemic stroke within 2 weeks
* Participants in whom one stent can't cover the lesion length or the use of multiple stents is required
* Greater than (>) 50% stenosis proximal or distal to the target intracranial lesion
* Intracranial arterial stenosis related to non-atherosclerotic factors, such as: arterial dissection, moya-moya disease; vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebrospinal fluid pleocytosis; radiation-induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; postpartum angiopathy; suspected vasospastic process, and developmental or genetic abnormalities
* Participants with symptoms of cerebral ischemia caused by cardiac embolism
* Severe vascular tortuosity, highly calcified or anatomy that would preclude the safe introduction of a guiding catheter, guiding sheath or stent placement
* Myocardial infarction within previous 30 days
* Permanent atrial fibrillation, persistent atrial fibrillation, any episode of paroxysmal atrial fibrillation within the past six months, or history of paroxysmal atrial fibrillation requiring chronic anticoagulation
* Intolerance or allergic reaction to any of antithrombotic therapy or medicine used during the procedure
* History of life-threatening allergy to contrast medium. If not life threatening and can be effectively pre-treated, participant can be enrolled at investigators' discretion
* Surgery within previous 30 days or planned in the next 90 days after enrollment
* Intracranial hemorrhage within 3 months
* Concomitant intracranial tumor, aneurysm or arteriovenous malformation
* Haemoglobin <10 grams per deciliter (g/dL), blood platelet count <80000 per milliliters (/ml), international normalization ratio >1.5, or other uncorrectable coagulopathies.
* Life expectancy of <3 years due to the concomitant illness.
* Pregnant or lactating women
* Participants judged unsuitable for stenting and angioplasty by the investigator

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with In-Stent Restenosis | At 12 months post-procedure
  In-stent restenosis greater than (>) 50 percent (%) at 12 months post-procedure as assessed by an independent Imaging Core Lab will be reported. The percent stenosis of an intracranial artery is calculated according to the warfarin-aspirin symptomatic intracranial disease (WASID) criteria: percent stenosis= ([1-{Dstenosis/Dnormal}]) * 100, where Dstenosis = the diameter of the artery at the site of the most severe stenosis and Dnormal = the diameter of the proximal normal artery.

SECONDARY OUTCOMES:
Number of Participants with Technical Success | Immediately post-procedure (Day 0)
  Technical success immediately post-procedure is defined as complete stent coverage and residual stenosis less than or equal to (<=) 50% as assessed by an independent Imaging Core Lab.
Number of Participants with In-Stent Restenosis | At 6 months post-procedure
  In-stent restenosis (>50%) at 6 months post-procedure as assessed by an independent Imaging Core Lab will be reported. The percent stenosis of an intracranial artery is calculated according to the warfarin-aspirin symptomatic intracranial disease (WASID) criteria: percent stenosis=([1-{Dstenosis/Dnormal}]) * 100, where Dstenosis = the diameter of the artery at the site of the most severe stenosis and Dnormal = the diameter of the proximal normal artery.
National Institutes of Health Stroke Scale (NIHSS) Scores | At 6 months and 12 months post-procedure
  NIHSS scores at 6 months and 12 months post-procedure will be reported. NIHSS score is a tool used to objectively quantify the impairment caused by a stroke and to evaluate stroke severity. It ranges from 0 to 42, with 42 being the highest and 0 being the lowest. The higher the NIHSS score, the worse the neurological function.
Modified Rankin Scale (mRS) Scores | At 30 days, 6 months and 12 months post-procedure
  mRS scores at 30 days, 6 months and 12 months post-procedure will be reported. mRS score is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke. It ranges from 0 to 5. The higher the mRS score, the worse the prognosis.
Number of Participants Free of Ischemic Stroke within the Territory of Stented Vessel | From 30 days to 12 months post-procedure
  Ischemic stroke within the territory of stented vessel from 30 days to 12 months post-procedure as assessed by the independent clinical events committee will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medos International SARL Clinical Trial, Study Director — Medos International SARL
Locations (14):
- China (14):
  - Xuanwu Hospital, Capital Medical University, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Haikou People's Hospital, Haikou
  - First Affiliated Hospital, Harbin Medical University, Harbin
  - Central Hospital Affiliated to Shandong First Medical University (Jinan Central Hospital), Jinan
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Provincial Hospital, Jinan
  - Nanjing Drum Tower Hospital, Nanjing
  - Ningbo First Hospital, Ningbo
  - Huashan Hospital Fudan University, Shanghai
  - Wenzhou Central Hospital, Wenzhou
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Redon J, Olsen MH, Cooper RS, Zurriaga O, Martinez-Beneito MA, Laurent S, Cifkova R, Coca A, Mancia G. Stroke mortality and trends from 1990 to 2006 in 39 countries from Europe and Central Asia: implications for control of high blood pressure. Eur Heart J. 2011 Jun;32(11):1424-31. doi: 10.1093/eurheartj/ehr045. Epub 2011 Apr 12. PMID 21487117
- [Background] Wong KS, Li H, Lam WW, Chan YL, Kay R. Progression of middle cerebral artery occlusive disease and its relationship with further vascular events after stroke. Stroke. 2002 Feb;33(2):532-6. doi: 10.1161/hs0202.102602. PMID 11823665
- [Background] Kasner SE, Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Benesch CG, Sila CA, Jovin TG, Romano JG, Cloft HJ; Warfarin Aspirin Symptomatic Intracranial Disease Trial Investigators. Predictors of ischemic stroke in the territory of a symptomatic intracranial arterial stenosis. Circulation. 2006 Jan 31;113(4):555-63. doi: 10.1161/CIRCULATIONAHA.105.578229. Epub 2006 Jan 23. PMID 16432056
- [Background] Famakin BM, Chimowitz MI, Lynn MJ, Stern BJ, George MG; WASID Trial Investigators. Causes and severity of ischemic stroke in patients with symptomatic intracranial arterial stenosis. Stroke. 2009 Jun;40(6):1999-2003. doi: 10.1161/STROKEAHA.108.546150. Epub 2009 Apr 30. PMID 19407228
- [Background] Fiorella D. Endovascular treatment of intracranial stenosis. World Neurosurg. 2011 Dec;76(6 Suppl):S66-70. doi: 10.1016/j.wneu.2011.07.024. PMID 22182273
- [Background] Bose A, Hartmann M, Henkes H, Liu HM, Teng MM, Szikora I, Berlis A, Reul J, Yu SC, Forsting M, Lui M, Lim W, Sit SP. A novel, self-expanding, nitinol stent in medically refractory intracranial atherosclerotic stenoses: the Wingspan study. Stroke. 2007 May;38(5):1531-7. doi: 10.1161/STROKEAHA.106.477711. Epub 2007 Mar 29. PMID 17395864
- [Background] Zaidat OO, Klucznik R, Alexander MJ, Chaloupka J, Lutsep H, Barnwell S, Mawad M, Lane B, Lynn MJ, Chimowitz M; NIH Multi-center Wingspan Intracranial Stent Registry Study Group. The NIH registry on use of the Wingspan stent for symptomatic 70-99% intracranial arterial stenosis. Neurology. 2008 Apr 22;70(17):1518-24. doi: 10.1212/01.wnl.0000306308.08229.a3. Epub 2008 Jan 30. PMID 18235078
- [Background] Fiorella DJ, Turk AS, Levy EI, Pride GL Jr, Woo HH, Albuquerque FC, Welch BG, Niemann DB, Aagaard-Kienitz B, Rasmussen PA, Hopkins LN, Masaryk TJ, McDougall CG. U.S. Wingspan Registry: 12-month follow-up results. Stroke. 2011 Jul;42(7):1976-81. doi: 10.1161/STROKEAHA.111.613877. Epub 2011 Jun 2. PMID 21636812
- [Background] Barnard ZR, Alexander MJ. Update in the treatment of intracranial atherosclerotic disease. Stroke Vasc Neurol. 2019 Oct 16;5(1):59-64. doi: 10.1136/svn-2019-000279. eCollection 2020. PMID 32411409
- [Background] Nordmeyer H, Chapot R, Haage P. Endovascular Treatment of Intracranial Atherosclerotic Stenosis. Rofo. 2019 Jul;191(7):643-652. doi: 10.1055/a-0855-4298. Epub 2019 Apr 4. English, German. PMID 30947351
- [Background] Tarabishy (2019). Counseling and Management of Patients with Intracranial Atherosclerosis Disease. In: Spiotta A., Turner R., Chaudry M., Turk A. (eds) Management of Cerebrovascular Disorders.
- [Background] Hurford R, Wolters FJ, Li L, Lau KK, Kuker W, Rothwell PM. Prognosis of Asymptomatic Intracranial Stenosis in Patients With Transient Ischemic Attack and Minor Stroke. JAMA Neurol. 2020 Aug 1;77(8):947-954. doi: 10.1001/jamaneurol.2020.1326. PMID 32453401
- [Background] Zhang Q, Dong K, Song H. Comparison of stent versus medical therapy for symptomatic patients with intracranial atherosclerotic stenosis: A meta-analysis. J Neurol Sci. 2017 Jan 15;372:272-278. doi: 10.1016/j.jns.2016.11.064. Epub 2016 Nov 25. PMID 28017227
- [Background] Krasteva MP, Lau KK, Mordasini P, Tsang ACO, Heldner MR. Intracranial Atherosclerotic Stenoses: Pathophysiology, Epidemiology, Risk Factors and Current Therapy Options. Adv Ther. 2020 May;37(5):1829-1865. doi: 10.1007/s12325-020-01291-4. Epub 2020 Apr 8. PMID 32270364
- [Background] Samuels OB, Joseph GJ, Lynn MJ, Smith HA, Chimowitz MI. A standardized method for measuring intracranial arterial stenosis. AJNR Am J Neuroradiol. 2000 Apr;21(4):643-6. PMID 10782772
- [Background] Chimowitz MI, Lynn MJ, Turan TN, Fiorella D, Lane BF, Janis S, Derdeyn CP; SAMMPRIS Investigators. Design of the stenting and aggressive medical management for preventing recurrent stroke in intracranial stenosis trial. J Stroke Cerebrovasc Dis. 2011 Jul-Aug;20(4):357-68. doi: 10.1016/j.jstrokecerebrovasdis.2011.05.001. PMID 21729789
- [Background] Bai WX, Gao BL, Li TX, Wang ZL, Cai DY, Zhu LF, Xue JY, Li ZS. Wingspan stenting can effectively prevent long-term strokes for patients with severe symptomatic atherosclerotic basilar stenosis. Interv Neuroradiol. 2016 Jun;22(3):318-24. doi: 10.1177/1591019915623797. Epub 2016 Jan 27. PMID 26823331
- [Background] Zhang Y, Rajah GB, Liu P, Sun Y, Liu T, Li X, Miao Z, Li G. Balloon-mounted versus self-expanding stents for symptomatic intracranial vertebrobasilar artery stenosis combined with poor collaterals. Neurol Res. 2019 Aug;41(8):704-713. doi: 10.1080/01616412.2019.1610837. Epub 2019 Apr 28. PMID 31030623
- [Background] Wang ZL, Gao BL, Li TX, Cai DY, Zhu LF, Xue JY, Bai WX, Li ZS. Outcomes of middle cerebral artery angioplasty and stenting with Wingspan at a high-volume center. Neuroradiology. 2016 Feb;58(2):161-9. doi: 10.1007/s00234-015-1611-8. Epub 2015 Oct 29. PMID 26515072
- [Background] Wang ZL, Gao BL, Li TX, Cai DY, Zhu LF, Bai WX, Xue JY, Li ZS. Symptomatic intracranial vertebral artery atherosclerotic stenosis (>/=70%) with concurrent contralateral vertebral atherosclerotic diseases in 88 patients treated with the intracranial stenting. Eur J Radiol. 2015 Sep;84(9):1801-4. doi: 10.1016/j.ejrad.2015.05.033. Epub 2015 Jun 5. PMID 26119803
- [Background] Gruber P, Garcia-Esperon C, Berberat J, Kahles T, Hlavica M, Anon J, Diepers M, Nedeltchev K, Remonda L. Neuro Elutax SV drug-eluting balloon versus Wingspan stent system in symptomatic intracranial high-grade stenosis: a single-center experience. J Neurointerv Surg. 2018 Dec;10(12):e32. doi: 10.1136/neurintsurg-2017-013699. Epub 2018 Apr 7. PMID 29627786
- [Background] Li TX, Gao BL, Cai DY, Wang ZL, Zhu LF, Xue JY, Bai WX, He YK, Li L. Wingspan Stenting for Severe Symptomatic Intracranial Atherosclerotic Stenosis in 433 Patients Treated at a Single Medical Center. PLoS One. 2015 Sep 30;10(9):e0139377. doi: 10.1371/journal.pone.0139377. eCollection 2015. PMID 26422692
- [Background] Ma N, Zhang Y, Shuai J, Jiang C, Zhu Q, Chen K, Liu L, Li B, Shi X, Gao L, Liu Y, Wang F, Li Y, Liu T, Zheng H, Mo D, Gao F, Wang Y, Wang Y, Feng L, Miao Z. Stenting for symptomatic intracranial arterial stenosis in China: 1-year outcome of a multicentre registry study. Stroke Vasc Neurol. 2018 May 7;3(3):176-184. doi: 10.1136/svn-2017-000137. eCollection 2018 Sep. PMID 30294474
- [Background] Lee KY, Chen DY, Hsu HL, Chen CJ, Tseng YC. Undersized angioplasty and stenting of symptomatic intracranial tight stenosis with Enterprise: Evaluation of clinical and vascular outcome. Interv Neuroradiol. 2016 Apr;22(2):187-95. doi: 10.1177/1591019915609165. Epub 2015 Nov 4. PMID 26542728
- [Background] Vajda Z, Schmid E, Guthe T, Klotzsch C, Lindner A, Niehaus L, Sperber W, Peters J, Arnold G, Bazner H, Henkes H. The modified Bose method for the endovascular treatment of intracranial atherosclerotic arterial stenoses using the Enterprise stent. Neurosurgery. 2012 Jan;70(1):91-101; discussion 101. doi: 10.1227/NEU.0b013e31822dff0f. PMID 21778921
- [Background] Wang X, Wang Z, Ji Y, Ding X, Zang Y, Wang C. Enterprise stent in recanalizing non-acute atherosclerotic intracranial internal carotid artery occlusion. Clin Neurol Neurosurg. 2017 Nov;162:47-52. doi: 10.1016/j.clineuro.2017.06.015. Epub 2017 Jun 27. PMID 28926782
- [Background] Salik AE, Selcuk HH, Zalov H, Kilinc F, Cirak M, Kara B. Medium-term results of undersized angioplasty and stenting for symptomatic high-grade intracranial atherosclerotic stenosis with Enterprise. Interv Neuroradiol. 2019 Oct;25(5):484-490. doi: 10.1177/1591019919832244. Epub 2019 Apr 16. PMID 30991867
- [Background] Qiu, X.,Ding, Y.,Xia, S.,Li, W.,Chen, L.,Xia, X.,Ke, S.,Wei, J.,Li, Q.,Peng, Z.. Effect evaluation of Enterprise stents in the treatment of complex and severe symptomatic intracranial atherosclerotic stenosis. Chinese Journal of Cerebrovascular Diseases. 2019. 16 (5):257-262
- [Background] Rubin, D.B., Multiple Imputation after 18+ Years. Journal of the American Statistical Association, 1996. 91(434): p. 473-489.